CLINICAL TRIAL: NCT03150888
Title: Multi-provincial Cohort for Hypertension in China
Brief Title: Multi-provincial Cohort for Hypertension (MUCH)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other); Beijing Tiantan Hospital (Other); Ruijin Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Southwest Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC0900902
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents; Heart Disease Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, blood cell, urine and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital based hypertension cohort
  Interventions: Drug: Antihypertensive Agents; Other: Cardiovascular risk factors
- Community based hypertension cohort
  Interventions: Drug: Antihypertensive Agents; Other: Cardiovascular risk factors

INTERVENTIONS:
Drug: Antihypertensive Agents — Single or combination therapy with five type of antihypertensive agents, such as Ca channel blockers, ACE inhibitors, ARBs, diuretics, or beta-blockers.
Other: Cardiovascular risk factors — Different level of cardiovascular risk factors associated with genetics, environments and lifestyles.

SUMMARY:
The purpose of this study is to construct hypertension specialized cohort using uniform standards and specifications. This study timely collected multi-dimensional clinical information through electronic medical records, mobile health, data integration, informatics and computer modern techniques, linking self-reported data and big data platforms from different sources to timely obtain the incidence and mortality data, and integrating hypertension cohort samples and the associated clinical records systematically, in order to build a 30-thousand hypertension specialized cohort with fine phenotypic data and blood/urine samples, thus far to provide support for the development of precise medicine research and related industries.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* over 18 years old
* ti sign the informed consent

Exclusion Criteria:

* with life-threatening severe disease, such as severe tumor or AIDs
* pregnancy or lactating women,or plan to pregnant within half a year,
* with severe mental disorders
* participating in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, and community sample
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Composite end point of major cardiovascular and cerebrovascular events | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 year
  Composite end point of major cardiovascular and cerebrovascular events

SECONDARY OUTCOMES:
New-onset of cardiovascular events | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 year
  New-onset of cardiovascular events
New-onset of stroke | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 year
  New-onset of stroke
Total death | From date of enrollment until date of death from all cause, assessed up to 3 year
  Total death
Major bleeding | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 year
  Major bleeding
Atrial fibrillation | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 year
  Atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, MD,PhD, Principal Investigator — Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Tiantan Hospital, Beijing
  - Beijing Tsinghua Chang Gung Hospital, Beijing
  - Southwest Hospital, China, Chongqing
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Ruijin Hospital, Shanghai